CLINICAL TRIAL: NCT05326451
Title: Home-based Transcranial Direct Current Stimulation Open Trial for Behavioral and Cognitive Symptoms in Huntington's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Erin Furr Stimming, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-1065
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Huntington Disease
Keywords: transcranial direct current stimulation
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- active tDCS (Experimental)
  Interventions: Device: active tDCS

INTERVENTIONS:
Device: active tDCS — Participants will receive active tDCS with a constant current intensity of 2mA. Anodal tDCS will be applied to the left dorsolateral prefrontal cortex, while cathodal electrode will be positioned on the right dorsolateral prefrontal cortex. Caregivers will help setting up and administering tDCS for participants with HD at home. tDCS will be applied for 30min at an intensity of 2mA, with 30 s ramping up and down. Sessions will be remotely supervised by trained research staff (RA), and will run from Monday through Friday for four consecutive weeks.

SUMMARY:
The purpose of this study is to assess feasibility, acceptability, and safety of providing transcranial direct current stimulation( tDCS) to Huntingtons Disease (HD) patients in the early to middle stages and to assess the efficacy of tDCS for HD-related behavioral, cognitive and other symptoms

ELIGIBILITY:
Participant:

Inclusion Criteria:

* confirmed HD mutation carriers and/or established family history alongside typical symptoms (i.e. chorea) of HD;
* early (stages 1 and 2) or moderate (stage 3) stages according to Shoulson-Fahn
* exhibit mild to moderate behavioral symptoms defined by severity scores in the PBA-S between 1 and 3 for any of the evaluated symptoms and no symptoms with a severity score of 4
* stable doses of medications for at least one month
* Have a caregiver willing to be present during tDCS sessions and answer questionnaires.

Exclusion Criteria:

* unstable medical conditions
* history of epilepsy
* metallic objects in the brain
* Have a caregiver willing to be present during tDCS sessions and answer questionnaires.
* clinical diagnosis of major cognitive disorder or dementia
* Have risk of suicidal behavior, defined as any suicidal behavior or suicidal ideation of type 4 or type 5 based on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the 3 months prior to screening
* simultaneous participation in other clinical trial
* Individuals determined to be incapable of consent per past medical history or via assessment by the study staff at time of consent.

Caregiver:

Inclusion Criteria:

-willingness to participate in the study

Exclusion Criteria:

-motor/cognitive symptoms related to Alzheimer's disease or Huntington's disease that might impair the ability to assist the participant during the research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by the number of participants included and who successfully completed the protocol | through study completion, an average of 8 weeks
Change in acceptability of the treatment as assessed by the tDCS acceptability questionnaire | Baseline, week 2, week 4, week 8
  Acceptability will be evaluated using a Likert scale (from 0 [strongly disagree] to 10 [strongly agree]) to answer ten affirmatives regarding the use of home based tDCS, with a total score range of 0-10 and a higher score indicating higher acceptability.
Change in safety of home-based tDCS treatment as as assessed by the tDCS side effect questionnaire | week 2, week 4
  Safety will be assessed with a 10-item questionnaire about side effects, including itching, burning, headache, fatigue, and dizziness. Each question is scored form 0-10, with a total score range of 0-10 and a higher score indicating more side effects.

SECONDARY OUTCOMES:
Change in Motor function as assessed by the Unified Huntington Disease Rating Scale (UHDRS) | Baseline,week4
  The motor section of the UHDRS consists of 31 items rated on a 5-point ordinal scale ranging from 0 to 4, with a score of 0 indicating no abnormalities and 4 indicating the most severe impairment. Total score range is 0 to 124, with a higher score indicating decreased inability to perform motor tasks.
Change in Cognitive function as assessed by the Unified Huntington Disease Rating Scale (UHDRS) | Baseline,week4
  The cognitive function section of the UHDRS consists of 5 items rated on a 5-point ordinal scale ranging from 0- to 4, with a total score range of 0 to 20 and with a higher score indicating better cognitive performance.
Change in Behavior as assessed by the Unified Huntington Disease Rating Scale (UHDRS) | Baseline,week4
  The behavioral section of the UHDRS consists of 11 items evaluating various behavioral signs and symptoms. Individuals are ranked on both severity and frequency on a 0 to 4 scale, with 0 being not present and 4 being severe and frequent. Total behavioral scores are calculated by summing the severity and frequency items, with a total score range of 0 (no behavioral symptoms) to 88 (most severe behavioral symptoms).
Change in apathy as assessed by the Brief Dimensional Apathy Scale (bDAS) | Baseline, week 2, week 4, week 8
  This scale consists of 9 questions, each scored from 0 (almost always) to 3 (hardly ever), with a total score range of 0 to 27 and a higher score indicating more apathy.
Change in depression as assessed by the Patient Health Questionnaire (PHQ-9) | Baseline, week 2, week 4, week 8
  This questionnaire has 9 questions. with each scored form 0 (not at all) to 3 (nearly every day), with a total score range of 0 to 27 and a higher score indicating more depression.
Change in irritability as assessed by the Irritability Questionnaire | Baseline, week 2, week 4, week 8
  This is a 21-item questionnaire, with each item scored form 0 (never) to 3 (most of the time), for a total score range of of 0 to 63 and a higher score indicating more irritability.
Change in cognition as assessed by the Montreal Cognitive Assessment (MoCA) | Baseline, week 2, week 4, week 8
  MoCA is scored from 0 to 30, with a higher score indicating better performance.
Change in anxiety and depressive symptoms as assessed by the Hospital Anxiety and Depression Scale (HADS) | Baseline, week 2, week 4, week 8
  HADS is a 14-item scale, with seven items each for anxiety and depression subscales. Scoring for each item ranges from 0 to 3, with a total score range of 0 to 42 and a total subscale score range of 0 to 21. A subscale score greater than 8 denotes anxiety or depression.
Change in behavioral symptoms as assessed by the Problem Behaviours Assessment (PBA-s) | Baseline, 2 weeks of treatment, at the end of treatment (week 4) and 4 weeks post-treatment.
  Each symptom is rated for severity on a 5-point scale : 0 = not at all; 1 = trivial; 2 = mild; 3 = moderate (disrupting everyday activities); and 4 = severe or intolerable. Each symptom is also scored for frequency on a 5-point scale as follows: 0 = symptom absent; 1 = less than once weekly; 2 = at least once a week; 3 = most days (up to and including some part of everyday); and 4 = all day, every day. Severity and frequency scores are multiplied to produce an overall 'PBA score' for each symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Stimming, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No